CLINICAL TRIAL: NCT02550795
Title: Effects of Single Dose Dexmedetomidine or Dexmedetomidine Combined With Dexamethasone on Postoperative Nausea and Vomiting in Breast Cancer
Brief Title: Dexmedetomidine or Dexmedetomidine Combined With Dexamethasone on Postoperative Nausea and Vomiting in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Breast PONV; GCIRB2014 (Registry Identifier: GCIRB2014-154)
Record Dates: First submitted 2015-08-30; First posted 2015-09-16 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): administration of 0.9% normal saline 10ml
  Interventions: Drug: Control
- Dexmedetomidine (Active Comparator): administration of 0.5ug/kg of dexmedetomidine (5ml)
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine and dexamethasone (Active Comparator): administration of 0.5 ug/kg of dexmedetomidine and dexamethasone 5mg (total 5ml)
  Interventions: Drug: Dexmedetomidine and dexamethasone

INTERVENTIONS:
Drug: Dexmedetomidine — administration of dexmedetomidine only
  Other Names: DO
  Arms: Dexmedetomidine
Drug: Dexmedetomidine and dexamethasone — administration of dexmedetomidine and dexamethasone
  Other Names: DD
  Arms: Dexmedetomidine and dexamethasone
Drug: Control — administration of normal saline
  Other Names: OO
  Arms: Control

SUMMARY:
Previous reports demonstrated that dexmedetomidine could reduce the incidence of postoperative nausea and vomiting (PONV). Dexamethason also had been commonly used for ajuvant drugs for preventing and reducing PONV. So investigator want to study about the effect of dexmedetomidine only or combined with dexamethasone for preventing PONV.

DETAILED DESCRIPTION:
Previous reports demonstrated that dexmedetomidine, a alpha 2 selective agonist could reduce the incidence of postoperative nausea and vomiting (PONV). Dexamethason also had been commonly used for ajuvant drugs for preventing and reducing PONV. So investigator want to study about the effect of dexmedetomidine only or combined with dexamethasone for preventing PONV.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical status I or II female scheduled for breast conserving surgery of modified radical mastectomy.

Exclusion Criteria:

* uncontrolled cardiovascular disease
* history of chronic pain
* smoker
* previous history of steroid administraion
* neoajuvant chemotherapy

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no one who excluded before assignment to groups
Period: Overall Study
Arm/Group | Control | Dexmedetomidine | Dexmedetomidine and Dexamethasone
Started | 50 | 50 | 50
Completed | 50 | 49 | 50
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Dexmedetomidine | Dexmedetomidine and Dexamethasone | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: one patient excluded from the analysis according to changes of surgery method
  years
    number analyzed (Participants) | 50 | 49 | 50 | 149
    (all) | 48.7 (6.4) | 48.2 (7.1) | 48.4 (7.5) | 48.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 50 | 150
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Nausea (Numeric Rating Scale for Nausea)
Description: Numeric rating scale for postoperative nausea (scores on a scale) (0-no symptoms; 10-worst symptoms imaginable). Ramosetron 0.3 mg was administered to patients with nausea >5 points on the numeric rating scale
Time Frame: Changes from baseline in postoperative nausea at 30 min
Population: Patients who underwent breast cancer surgery
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Control | Dexmedetomidine | Dexmedetomidine and Dexamethasone
Number analyzed (Participants) | 50 | 49 | 50
scores on a scale | 0 [0 to 0.25] | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: Postoperative Vomiting (Number of Participants With Vomiting)
Description: frequencies of vomiting (number of participants with vomiting) 24 hour post-operatively
Time Frame: Changes from baseline in postoperative nausea at 30 min
Population: Patients who underwent breast cancer surgery
Measure: Number; unit: participants
Arm/Group | Control | Dexmedetomidine | Dexmedetomidine and Dexamethasone
Number analyzed (Participants) | 50 | 49 | 50
participants
  0-1 hour | 4 | 0 | 0
  1-6 hour | 15 | 6 | 1
  6-24hour | 9 | 5 | 1

3. Secondary Outcome: Rhodes Index Score
Description: Rhodes Index of nausea, vomiting, and retching at 6 to 24 hours after surgery (ask 8 question about discomfort due to PONV and each questions are consist of 0~4 score) (minimal PONV 0 to maximal PONV 32) lower values represent a bettwer outcome
Time Frame: assessed at 6 and 24 hour after operative end
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Dexmedetomidine | Dexmedetomidine and Dexamethasone
Number analyzed (Participants) | 50 | 49 | 50
score on a scale
  1-6 hour after surgery | 5 [0 to 12] | 0 [0 to 5.5] | 0 [0 to 0.5]
  6-24 hour after surgery | 3.5 [0 to 13] | 0 [0 to 3.5] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Control | Dexmedetomidine | Dexmedetomidine and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No